CLINICAL TRIAL: NCT01182532
Title: A Clinical Trial to Evaluate the Effectiveness and Safety of Chinese Medicine in the Treatment of Mild Type of Hand, Foot, and Mouth Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine (Other)
Collaborators: Beijing University of Chinese Medicine (Other); China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Guoliang Zhang, Chief, The First Affiliated Hospital of Anhui University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200907001-3
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-07

CONDITIONS: Hand, Foot and Mouth Disease
Keywords: Mild type of hand, foot and mouth disease; Traditional Chinese Medicine; Effectiveness; Safety
MeSH Terms: conditions — Hand, Foot and Mouth Disease; Mouth Diseases | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Western therapy (Active Comparator)
  Interventions: Other: Western therapy
- TCM treatment (Experimental)
  Interventions: Drug: TCM Syndrome Differentiation and Treatment
- Western therapy plus TCM treatment (Experimental): The combination of both western therapy and TCM treatment.
  Interventions: Other: Western therapy plus TCM treatment

INTERVENTIONS:
Other: Western therapy — Symptomatic treatment: vitamin B, vitamin C, mouth care and skin care.
  1. Adopting physical cooling therapy, including physical cooling paste or warm bathing, when patient's body temperature is lower than 38.5 degree Celsius;
  2. Using Ibuprofen suspension when patient's temperature higher than 38.5 degree Celsius;
  Arms: Western therapy
Drug: TCM Syndrome Differentiation and Treatment — 1. Lung-Spleen Damp-Heat Syndrome Symptoms: Fever, maculopapule and herpes on hand, foot and buttock; herpes on oral mucous membrane; redness in throat, salivation, tiredness, faint red tongue or reddish tongue, greasy fur, speedy pulse, red and purple fingerprint.
     Formula: Forsythia suspensa (Thunb.) vahl.(Lian Qiao), Lonicera japonica Thunb (Jin Yin Hua), Scutellaria baicalensis Georgi (Huang Qin), etc.
     Dosage: Adjusting by age and weight of patients. Decoction.
  2. Dampness-Heat Retention Syndrome Symptoms: High fever, dirty color of tetter, tiredness, oral ulcer, reddish tongue or deep red tongue, little saliva, yellow and greasy fur, fine and rapid pulse, deep purple fingerprint.
  Formula: Forsythia suspensa (Thunb.) vahl.(Lian Qiao), Gardenia jasminoides Ellis (rough Zhi Zi), Scutellaria baicalensis Georgi (Huang Qin), etc.
  Dosage: Adjusting by age and weight of patients. Decoction.
  Arms: TCM treatment
Other: Western therapy plus TCM treatment — 1. Symptomatic treatment using the same treatment methods in western therapy group;
  2. Syndrome differentiation and treatment adopting the same methods in TCM treatment group.
  Arms: Western therapy plus TCM treatment

SUMMARY:
The study is aimed to evaluate the effectiveness and safety of traditional Chinese medicine (TCM) for treatment of hand, foot, and mouth disease (HFMD).

DETAILED DESCRIPTION:
By adopting a multi-center, randomized and controlled clinical trial, this study is aimed to evaluate the effectiveness, safety and economic evaluation of traditional Chinese medicine for treatment of HFMD, and to provide scientific evidence for the construction of TCM methods in treating HFMD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of severe hand-foot-mouth disease patients according to Hand-Foot-Mouth Disease Treatment Guidelines 2010 issued by China's Ministry of Health; More than 1/3 patients should be diagnosed by etiological examination.
* Less than 48 hours of occurrence of fever and/or occurrence of tetter or herpes.
* Age of 1-14 years.
* Patients or their guardians agree to participate in this study and signed the informed consent form.

Exclusion Criteria:

* Complicated with other serious primary diseases in organ such as congenital heart disease, chronic hepatitis, nephritis and blood diseases, etc.
* With history of allergies on traditional Chinese medicine.
* Patients or their guardians suffering from Psychiatric diseases.
* Attending other clinical studies on HFMD after diagnosed.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3000 (Actual)
Dates: Start 2010-05; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
time to onset | 10 days
  Refering to the length of time to bring down the fever by 0.5 degrees Celsius after the medicine is taken.
time of body temperature going back to normal | 10 days
  Refering to the time of the armpit temperature of lower than 37.0 degrees Celsius, lasting for at least 24 hours, after the medicine is taken.

SECONDARY OUTCOMES:
time of symptom disappearance | 10 days
  Refering to the length of time when clinical symptoms and signs totally disappere after the medicine is used.
case severity rate | 10 days
  Refering to the ratio of patient with mild type of HFMD to severe type, such as damage of central nervous system, pulmonary edema, heart failure, respiratory failure, etc.
time of tetter and oral ulcer disappearance | 10 days
  Refering to the length of time when the tetter due to HFMD disappears, characterised by no new tetter and oral ulcer develops, scab(s) or dropping; and time of oral ulcer concrescence, etc.
direct medical cost | 10 days
  Referring to the costs in the treatment of HFMD and relative disease, including the registration fee, examination fee, and drug fees, etc.
safety outcome | 10 days
  Calculated by adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Guoliang Zhang, Principal Investigator — An'Hui Chinese Medical College Affiliated No.1 Hospital
Locations (21):
- China (21):
  - Anhui Provincial Children's Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui College of Traditional Chinese Medicine, Hefei, Anhui
  - Beijing Ditan Hospital, Beijing, Beijing Municipality
  - Beijing You-An Hospital, Beijing, Beijing Municipality
  - Chongqing Hospital of Traditional Chinese Medicine, Chongqing, Chongqing Municipality
  - Fuzhou Infectious Disease Hospital, Fuzhou, Fujian
  - Xiamen Hospital of Traditional Chinese Medicine, Xiamen, Fujian
  - First Hospital of Lanzhou University, Lanzhou, Gausu
  - Shenzhen Third People's Hospital, Shenzhen, Guangzhou
  - The Fifth Hospital of Shijiazhuang, Hebei, Shijiazhuang, Hebei
  - Wuhan Hospital for Infectious Diseases, Wuhan, Hubei
  - Huhehaote Second Hospital, Hohhot, Inner Mongolia
  - Ninth Hospital of Nanchang, Nanchang, Jiangxi
  - Changchun Infectious Diseases Hospital, Changchun, Jilin
  - Ningxia Hui Autonomous Region Forth People's Hospital, Yinchuan, Ningxia Hui Autonomous
  - The Eighth Hospital of Xi'an City, Xi'an, Shaanxi
  - Shanghai Public Health Center, Shanghai, Shanghai Municipality
  - Chengdu Hospital for Infectious Diseases, Chengdu, Sichuan
  - Xinjiang Hongxing Hospital, Urumuqi, Xinjiang
  - First Affiliated Hospital to Kunming Medical College, Kunming, Yunnan
  - The Sixth People's Hospital of Hangzhou, Hangzhou, Zhejiang